CLINICAL TRIAL: NCT02020499
Title: Non-interventional, Observational, Long Term Study to Evaluate Common Therapeutic Algorithms and Possible Predictive Parameters for Somatuline Autogel (ATG) Treatment in Patients With Acromegaly.
Brief Title: Predictive Factors Study
Acronym: TAPAS
Status: Terminated | Type: Observational
Why Stopped: Poor enrolment
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-9B-52030-265
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acromegalic patients: Acromegalic subjects treated with Somatuline Autogel® (Lanreotide)
  Interventions: Drug: Somatuline Autogel® (lanreotide) 60, 90, 120 mg.

INTERVENTIONS:
Drug: Somatuline Autogel® (lanreotide) 60, 90, 120 mg. — Patients receiving treatment as prescribed by the investigator and according to current treatment recommendations and routine clinical practice, and in line with local regulations.

SUMMARY:
This is a long term study to evaluate common therapeutic algorithms and possible predictive parameters for Somatuline Autogel treatment in patients with Acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acromegaly.
* Males and females aged 18 years and older.
* Signed informed consent (patient must give consent to the collection of retrospective data).
* Patients who have had surgery may enter the study 3 months post-surgery and evaluated for the duration of the study.
* With the intention to be treated with ATG (decision to prescribe ATG made prior to inclusion into the study) or already being treated with ATG.
* If already being treated with ATG:

Previous ATG treatment maximum of 3 months. AND Minimum data available (demographic data, disease history including previous treatments, GH, IGF-1 levels at baseline and under treatment as applicable).

* Not receiving Dopamine Agonists or other medical therapy (Pegvisomant, or other somatostatin analogues) for the treatment or symptom control of acromegaly.

Exclusion Criteria:

* The subject has had radiotherapy in the last 5 years.
* The subject has had surgery in the last 3 months.
* The subject has already been included in this study.
* Participation in an interventional trial, or receiving experimental drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects in hospitals and private practices, suffering from acromegaly who are scheduled to receive ATG or already on treatment with ATG for a maximum of 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Growth hormone (GH) and insulin-like growth factor-1 (IGF-1) levels from baseline | Baseline and 4 weeks

SECONDARY OUTCOMES:
Change in Growth hormone (GH) and insulin-like growth factor-1 (IGF-1) levels from baseline | Baseline, 1 year and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (6):
- Australia (6):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St Vincent's Hospital, Fitzroy, Victoria
  - The Austin Hospital, Heidelberg, Victoria